CLINICAL TRIAL: NCT02278120
Title: A Phase III Randomized, Double-blind, Placebo-controlled Study of LEE011 or Placebo in Combination With Tamoxifen and Goserelin or a Non-steroidal Aromatase Inhibitor (NSAI) and Goserelin for the Treatment of Premenopausal Women With Hormone Receptor Positive, HER2-negative, Advanced Breast Cancer
Brief Title: Study of Efficacy and Safety in Premenopausal Women With Hormone Receptor Positive, HER2-negative Advanced Breast Cancer
Acronym: MONALEESA-7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEE011E2301; 2014-001931-36 (EudraCT Number)
Record Dates: First submitted 2014-10-22; First posted 2014-10-29 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Advanced Metastatic Breast Cancer
Keywords: LEE011; ribociclib; HR-positive; HER2-negative; Advanced breast cancer; Letrozole; Anastrozole; Tamoxifen; Goserelin; CDK; CDK4; CDK6; CDK4/6; Phase III; ER-positive; PR-positive; Premenopausal
MeSH Terms: interventions — ribociclib; Tamoxifen; Letrozole; Anastrozole; Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib + NSAI/tamoxifen + goserelin (Experimental): Ribociclib 600 mg daily oral (3 weeks on/ 1 week off) in combination with NSAI or tamoxifen (tamoxifen 20 mg daily oral or letrozole 2.5 mg daily oral or anastrozole 1 mg daily oral) and goserelin 3.6 mg subcutaneous injection (once every 28 days)
  Interventions: Drug: Ribociclib; Drug: Tamoxifen; Drug: Letrozole; Drug: Anastrozole; Drug: Goserelin
- Placebo + NSAI/tamoxifen + goserelin (Placebo Comparator): Placebo daily oral (3 weeks on/ 1 week off) in combination with NSAI or tamoxifen (tamoxifen 20 mg daily oral or letrozole 2.5 mg daily oral or anastrozole 1 mg daily oral) and goserelin 3.6 mg subcutaneous injection (once every 28 days).
  Participants were unblinded once the final OS analysis was conducted and after the implementation of protocol amendment 6 (16-Jul-2019) and were given the option to crossover to treatment with ribociclib +NSAI/tamoxifen + goserelin.
  Interventions: Drug: Tamoxifen; Drug: Letrozole; Drug: Anastrozole; Drug: Goserelin; Drug: Placebo

INTERVENTIONS:
Drug: Ribociclib — Ribociclib (600 mg, in three 200 mg hard gelatin capsules) was administered orally once daily on Days 1-21 of each 28-day cycle.
  Other Names: LEE011
  Arms: Ribociclib + NSAI/tamoxifen + goserelin
Drug: Tamoxifen — Tamoxifen (20 mg, tablets) was administered orally on a continuous daily schedule (days 1-28 of each 28-day cycle)
Drug: Letrozole — Letrozole (2.5 mg, tablets) was administered orally once daily on a continuous daily schedule (days 1-28 of each 28-day cycle)
Drug: Anastrozole — Anastrozole (1 mg, tablets) was administered orally once daily on a continuous daily schedule (days 1-28 of each 28-day cycle)
Drug: Goserelin — Goserelin (3.6 mg, subcutaneous implant) was administered on day 1 of every 28-day cycle
Drug: Placebo — Placebo (hard gelatin capsules) was administered orally once daily on Days 1-21 of each 28-day cycle.
  Arms: Placebo + NSAI/tamoxifen + goserelin

SUMMARY:
The purpose of this study was to determine whether treatment with tamoxifen or a non-steroidal aromatase inhibitors (NSAI) + goserelin + LEE011 prolonged progression-free survival (PFS) compared to treatment with tamoxifen or a NSAI + goserelin + placebo in premenopausal women with hormone receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer.

DETAILED DESCRIPTION:
This was a randomized, Phase III, double-blind, global study comparing the treatment efficacy and safety of ribociclib + goserelin + tamoxifen or a NSAI (letrozole or anastrozole) versus placebo + goserelin + tamoxifen or a NSAI in premenopausal women with HR+, HER2- advanced breast cancer.

Eligible participants were randomized in a 1:1 ratio to either the ribociclib arm or the placebo arm. Study treatment continued until disease progression, unacceptable toxicity, death, or discontinuation for any other reason.

Participants who discontinued treatment due to reasons other than disease progression or withdrawal of consent for efficacy follow-up continued to be monitored until disease progression, death, withdrawal of consent, loss to follow-up, or subject/guardian decision (post-treatment efficacy follow-up).

All participants who discontinued treatment were followed for survival until the predetermined number of overall survival (OS) events was reached.

Following the final OS analysis (performed when approximately 189 deaths were recorded) and with protocol amendment 6 (dated 18-Jul-2019), participants and investigators were unblinded and those participants in the placebo arm had the opportunity to cross-over to the ribociclib arm to receive ribociclib + goserelin + NSAI. Cross-over was optional and was conducted at the investigator's discretion and upon participant consent.

ELIGIBILITY:
Key inclusion criteria:

* Patients had advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy
* Patients were premenopausal or perimenopausal at the time of study entry
* Patients who had received (neo) adjuvant therapy for breast cancer were eligible
* Patients had a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer
* Patients had HER2-negative breast cancer
* Patients must have either had measurable disease or If no measurable disease was present, then at least one predominantly lytic bone lesion
* Patients had an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients had adequate bone marrow and organ function

Key exclusion criteria:

* Patients who had received a prior CDK4/6 inhibitor
* Patients were postmenopausal
* Patients who currently had inflammatory breast cancer at screening.
* Patients who had received any prior hormonal anti-cancer therapy for advanced breast cancer, except for ≤ 14 days of tamoxifen or NSAI ± goserelin for advanced breast cancer prior to randomization.
* Patients had a concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated basal cell skin carcinoma, squamous cell skin carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Patients with CNS metastases.
* Patients had active cardiac disease or a history of cardiac dysfunction
* Patients were currently using other antineoplastic agents
* Patients were pregnant or nursing or physiologically capable of becoming pregnant and not using highly effective contraception.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 672 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (163):
- United States (35):
  - Comprehensive Blood and Cancer SC-2, Bakersfield, California
  - University Of California Los Angeles Dept of Onc, Los Angeles, California
  - Comprehensive Cancer Center at Saint Joseph Hospital SC, Denver, Colorado
  - Danbury Hospital SC, Danbury, Connecticut
  - Florida Cancer Specialists Onc Dept, Fort Myers, Florida
  - Florida Cancer Specialists SC-2, Fort Myers, Florida
  - Memorial Cancer Institute SC, Hollywood, Florida
  - University Of Miami Univ Miami 2, Miami, Florida
  - NorthWest Georgia Oncology Centers IRB, Marietta, Georgia
  - Moanalua Medical Center. Attn: Oncology Dept SC, Honolulu, Hawaii
  - University of Chicago SC-3, Chicago, Illinois
  - Norton Cancer Institute SC, Louisville, Kentucky
  - Sidney Kimmel CCC At JH Dept of Onc., Baltimore, Maryland
  - Massachusetts General Hospital Onc Dept, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Onc Dept, Ann Arbor, Michigan
  - Washington Uni School of Med SC, St Louis, Missouri
  - Meridian Health Systems SC, Neptune City, New Jersey
  - University of New Mexico Hospital SC-2, Albuquerque, New Mexico
  - Clinical Research Alliance ., Lake Success, New York
  - Duke Univ Medical Center Duke (SC), Durham, North Carolina
  - Penn State University Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Bon Secours Cancer Center SC, Greenville, South Carolina
  - Erlanger Medical Center SC, Chattanooga, Tennessee
  - SCRI Oncology Partners Tennessee Oncology (3), Nashville, Tennessee
  - The Center for Cancer and Blood Disorders SC, Fort Worth, Texas
  - Methodist Hospita Methodist Can Cen Dept of Oncology, Houston, Texas
  - Uni of TX MD Anderson Cancer Cntr SC-5, Houston, Texas
  - Mays Cancer Ctr Uthsa Mdacc SC-4, San Antonio, Texas
  - Brooke Army Medical Center SC, San Antonio, Texas
  - Northern Utah Cancer Associates, Ogden, Utah
  - Bon Secours Virginia Health System, Midlothian, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Kadlec Clinic Hematology and Onco Kadlec Clinic Hematology & Onc, Kennewick, Washington
  - Northwest Medical Specialties Dept of Onc, Tacoma, Washington
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Univ Wisc 3, Madison, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, San Salvador de Jujuy, Jujuy Province
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, La Rioja
- Australia (5):
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Wilrijk
- Brazil (5):
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Passo Fundo, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Colombia (2):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Montería
- France (8):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (12):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Ulm
- Greece (2):
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Heraklion Crete
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Wan Chai
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szolnok
- India (4):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Mumbai
- Italy (20):
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Benevento, BN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Lucca, LU
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Napoli
- Lebanon (4):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Malaysia (2):
  - Novartis Investigative Site, Johor Bahru, Johor
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (3):
  - Novartis Investigative Site, Metepec, Edo. de México
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Monterrey Nuevo Leon, Monterrey
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Konin
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (2):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul
- Spain (14):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Geneva, Switzerland
- Taiwan (5):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Diyarbakır
  - Novartis Investigative Site, Edirne
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Al Ain Abu Dhabi, United Arab Emirates, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hart LL, Im SA, Tolaney SM, Campone M, Pluard T, Sousa B, Freyer G, Decker T, Kalinsky K, Sopher G, Gao M, Hu H, Kuemmel S. Efficacy, safety, and patient-reported outcomes across young to older age groups of patients with HR+/HER2- advanced breast cancer treated with ribociclib plus endocrine therapy in the randomized MONALEESA-2, -3, and -7 trials. Eur J Cancer. 2025 Feb 25;217:115225. doi: 10.1016/j.ejca.2025.115225. Epub 2025 Jan 8. PMID 39826197
- [Derived] Andre F, Su F, Solovieff N, Hortobagyi G, Chia S, Neven P, Bardia A, Tripathy D, Lu YS, Lteif A, Taran T, Babbar N, Slamon D, Arteaga CL. Pooled ctDNA analysis of MONALEESA phase III advanced breast cancer trials. Ann Oncol. 2023 Nov;34(11):1003-1014. doi: 10.1016/j.annonc.2023.08.011. Epub 2023 Sep 5. PMID 37673211
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111
- [Derived] Lu YS, Im SA, Colleoni M, Franke F, Bardia A, Cardoso F, Harbeck N, Hurvitz S, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva Vazquez R, Jung KH, Babu KG, Wheatley-Price P, De Laurentiis M, Im YH, Kuemmel S, El-Saghir N, O'Regan R, Gasch C, Solovieff N, Wang C, Wang Y, Chakravartty A, Ji Y, Tripathy D. Updated Overall Survival of Ribociclib plus Endocrine Therapy versus Endocrine Therapy Alone in Pre- and Perimenopausal Patients with HR+/HER2- Advanced Breast Cancer in MONALEESA-7: A Phase III Randomized Clinical Trial. Clin Cancer Res. 2022 Mar 1;28(5):851-859. doi: 10.1158/1078-0432.CCR-21-3032. PMID 34965945
- [Derived] Bardia A, Su F, Solovieff N, Im SA, Sohn J, Lee KS, Campos-Gomez S, Jung KH, Colleoni M, Vazquez RV, Franke F, Hurvitz S, Harbeck N, Chow L, Taran T, Rodriguez Lorenc K, Babbar N, Tripathy D, Lu YS. Genomic Profiling of Premenopausal HR+ and HER2- Metastatic Breast Cancer by Circulating Tumor DNA and Association of Genetic Alterations With Therapeutic Response to Endocrine Therapy and Ribociclib. JCO Precis Oncol. 2021 Sep 1;5:PO.20.00445. doi: 10.1200/PO.20.00445. eCollection 2021. PMID 34504990
- [Derived] Burris HA, Chan A, Bardia A, Thaddeus Beck J, Sohn J, Neven P, Tripathy D, Im SA, Chia S, Esteva FJ, Hart L, Zarate JP, Ridolfi A, Lorenc KR, Yardley DA. Safety and impact of dose reductions on efficacy in the randomised MONALEESA-2, -3 and -7 trials in hormone receptor-positive, HER2-negative advanced breast cancer. Br J Cancer. 2021 Aug;125(5):679-686. doi: 10.1038/s41416-021-01415-9. Epub 2021 Jun 22. PMID 34158598
- [Derived] Prat A, Chaudhury A, Solovieff N, Pare L, Martinez D, Chic N, Martinez-Saez O, Braso-Maristany F, Lteif A, Taran T, Babbar N, Su F. Correlative Biomarker Analysis of Intrinsic Subtypes and Efficacy Across the MONALEESA Phase III Studies. J Clin Oncol. 2021 May 1;39(13):1458-1467. doi: 10.1200/JCO.20.02977. Epub 2021 Mar 26. PMID 33769862
- [Derived] Yardley DA. MONALEESA clinical program: a review of ribociclib use in different clinical settings. Future Oncol. 2019 Aug;15(23):2673-2686. doi: 10.2217/fon-2019-0130. Epub 2019 Jul 15. PMID 31305131
- [Derived] Im SA, Lu YS, Bardia A, Harbeck N, Colleoni M, Franke F, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva-Vazquez R, Jung KH, Chakravartty A, Hughes G, Gounaris I, Rodriguez-Lorenc K, Taran T, Hurvitz S, Tripathy D. Overall Survival with Ribociclib plus Endocrine Therapy in Breast Cancer. N Engl J Med. 2019 Jul 25;381(4):307-316. doi: 10.1056/NEJMoa1903765. Epub 2019 Jun 4. PMID 31166679
- [Derived] Tripathy D, Im SA, Colleoni M, Franke F, Bardia A, Harbeck N, Hurvitz SA, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva Vazquez R, Jung KH, Babu KG, Wheatley-Price P, De Laurentiis M, Im YH, Kuemmel S, El-Saghir N, Liu MC, Carlson G, Hughes G, Diaz-Padilla I, Germa C, Hirawat S, Lu YS. Ribociclib plus endocrine therapy for premenopausal women with hormone-receptor-positive, advanced breast cancer (MONALEESA-7): a randomised phase 3 trial. Lancet Oncol. 2018 Jul;19(7):904-915. doi: 10.1016/S1470-2045(18)30292-4. Epub 2018 May 24. PMID 29804902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 185 sites across 30 countries.
Pre-assignment Details: Screening assessments were conducted up to 28 days prior to the randomization
Groups:
- Placebo + NSAI/Tamoxifen+ Goserelin: Placebo daily oral (3 weeks on/ 1 week off) in combination with NSAI or tamoxifen (tamoxifen 20 mg daily oral or letrozole 2.5 mg daily oral or anastrozole 1 mg daily oral) and goserelin 3.6 mg subcutaneous injection (once every 28 days).
  Participants were unblinded once the final OS analysis was conducted and after the implementation of protocol amendment 6 (16-Jul-2019) and were given the option to crossover to treatment with ribociclib +NSAI/tamoxifen + goserelin
Period: Treatment Period
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Started | 335 | 337
Crossover Cohort (Participants in the placebo arm who crossed over to the ribociclib arm and received at least one dose of the crossover study treatment) | 0 | 17
Completed | 0 | 0
Not Completed | 335 | 337
Not completed — Progressive disease | 234 | 260
Not completed — Subject/guardian decision | 23 | 20
Not completed — Adverse Event | 16 | 14
Not completed — Physician Decision | 14 | 27
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol deviation | 0 | 2
Not completed — Study terminated as per protocol | 43 | 11
Period: Post-treatment Efficacy Follow-up
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Started | 22 | 15
Completed | 0 | 1
Not Completed | 22 | 14
Not completed — Death | 0 | 1
Not completed — Subject/guardian decision | 1 | 2
Not completed — Study terminated as per protocol | 8 | 3
Not completed — Progressive disease | 12 | 7
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin | Total
Number analyzed (Participants) | 335 | 337 | 672
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (6.6) | 43.7 (6.17) | 43.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335 | 337 | 672
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 187 | 201 | 388
  Asian | 99 | 99 | 198
  Black | 10 | 9 | 19
  Native American | 3 | 3 | 6
  Other | 16 | 7 | 23
  Unknown | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Investigator Assessment
Description: PFS was defined as the period starting from the date of randomization to the date of the first documented progression or death caused by any reason. In cases where patients did not experience an event, the PFS was censored at the date of the last adequate tumor assessment. Clinical deterioration without objective radiological evidence was not considered as documented disease progression. PFS was assessed via local radiology assessment according to RECIST 1.1. As per protocol, the final PFS analysis was conducted after approximately 392 PFS events were documented. The Kaplan-Meier method was used to estimate PFS, and the median PFS, along with 95% confidence intervals, was reported for each treatment group. A stratified Cox regression model was used to estimate the hazard ratio of PFS, along with 95% confidence interval
Time Frame: From randomization to first documented progression or death, assessed up to approximately 29 months
Population: The Full Analysis Set (FAS) including all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo + NSAI/Tamoxifen+ Goserelin: Placebo daily oral (3 weeks on/ 1 week off) in combination with NSAI or tamoxifen (tamoxifen 20 mg daily oral or letrozole 2.5 mg daily oral or anastrozole 1 mg daily oral) and goserelin 3.6 mg subcutaneous injection (once every 28 days).
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Months | 23.8 [19.2 to NA] — NA = The value was not estimable due to insufficient number of participants with events | 13.0 [11.0 to 16.4]
Statistical Analysis 1: Comparison: Ribociclib + NSAI/Tamoxifen + Goserelin vs Placebo + NSAI/Tamoxifen+ Goserelin; Test type: Superiority; p < 0.0000001, Log Rank; Hazard Ratio, log = 0.553, 95% CI 2-sided [0.441 to 0.694]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. In cases where the patient's death was not recorded, the OS value was censored at the date of the last known patient's survival status. OS was estimated using the Kaplan-Meier method. As per protocol, the final OS analysis was conducted after approximately 189 deaths were documented.
  The median OS, along with 95% confidence intervals, was reported for each treatment group.The distribution of OS between the two treatment arms was compared using a log-rank test at one-sided cumulative 2.5% level of significance. A stratified Cox regression was used to estimate the OS hazard ratio and the associated 95% CI.
Time Frame: From randomization to death, assessed up to approximately 45 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Months | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | 40.9 [37.8 to NA] — NA: Not estimable due to the insufficient number of participants with events
Statistical Analysis 1: Comparison: Ribociclib + NSAI/Tamoxifen + Goserelin vs Placebo + NSAI/Tamoxifen+ Goserelin; Test type: Superiority; p = 0.00973, Log Rank — One-sided stratified log-rank test; Cox Proportional Hazard = 0.712, 95% CI 2-sided [0.535 to 0.948]

3. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment
Description: ORR is the percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 as per local assessment. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 29 months
Population: FAS including all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Percentage of participants | 40.9 [35.6 to 46.2] | 29.7 [24.8 to 34.6]
Statistical Analysis 1: Comparison: Ribociclib + NSAI/Tamoxifen + Goserelin vs Placebo + NSAI/Tamoxifen+ Goserelin; Test type: Superiority; p = 0.000980, Cochran-Mantel-Haenszel

4. Secondary Outcome: Clinical Benefit Rate (CBR) by Investigator Assessment
Description: Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1 and local assessment. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease: PD = At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20% the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to approximately 29 months
Population: FAS including all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Percentage of participants | 79.1 [74.8 to 83.5] | 69.7 [64.8 to 74.6]
Statistical Analysis 1: Comparison: Ribociclib + NSAI/Tamoxifen + Goserelin vs Placebo + NSAI/Tamoxifen+ Goserelin; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel

5. Secondary Outcome: Time to Response (TTR) by Investigator Assessment
Description: Time to response is the time from the date of randomization to the first documented response (CR or PR, which must be confirmed subsequently) according to RECIST 1.1 as per local assessment. The Kaplan-Meier method was used to estimate TTR, and the median TTR, along with 95% confidence intervals, was reported for each treatment group. Participants who did not achieve a confirmed response were censored at the maximum follow-up time for patients who had a PFS event (i.e. either progressed or died due to any cause) or at the date of last adequate tumor assessment otherwise.
  CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 29 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
months | NA [NA to NA] — N/A = The values were not evaluable due to insufficient number of participants with events | NA [NA to NA] — N/A = The values were not evaluable due to insufficient number of participants with events

6. Secondary Outcome: Duration of Response (DOR) by Investigator Assessment
Description: DOR was defined as the time from the first documented response (CR or PR) to the first documented progression or death due to underlying cancer as defined in RECIST 1.1 per investigator assessment. The Kaplan-Meier method was used to estimate DOR, and the median DOR, along with 95% confidence intervals, was reported for each treatment group. If a participant had not had an event, duration was censored at the date of last adequate tumor assessment.
  CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 29 months
Population: Randomized participants with confirmed CR or PR as per investigator assessment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 137 | 100
Months | 21.3 [18.3 to NA] — NA = The value was not estimable due to insufficient number of participants with events. | 17.5 [12.0 to NA] — NA = The value was not estimable due to insufficient number of participants with events.

7. Secondary Outcome: Time to Definitive Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) by at Least One Category of the Score
Description: ECOG PS categorized patients based on their ability to perform daily activities and self-care, with scores ranging from 0 to 5. A score of 0 indicated no restrictions in activity, while higher scores indicated increasing limitations. Time to definitive deterioration was defined as the time from the date of randomization to the date of the event, defined as experiencing an increase in ECOG PS by at least one category from the baseline or death. A deterioration was considered definitive if no improvements in the ECOG PS were observed at a subsequent time. The Kaplan-Meier method was used to estimate the distribution, and the median time to definitive deterioration, along with 95% confidence intervals, was reported for each treatment group. Patients receiving any further therapy prior to definitive worsening were censored at their date of last assessment prior to start of therapy. Patients that had not worsened at the data cutoff point were censored at the date of last assessment.
Time Frame: Baseline, up to approximately 29 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Months | NA [NA to NA] — NA = The value was not estimable due to insufficient number of participants with events | NA [NA to NA] — NA = The value was not estimable due to insufficient number of participants with events

8. Secondary Outcome: Time to Definitive 10% Deterioration in the Global Health Status/Quality of Life (GHS/QoL) Scale Score of the European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, 1 GHS/QoL scale, and 6 single items. GHS/QoL scale score ranges between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.The time to definitive 10% deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10% relative to baseline worsening of the QoL score (without further improvement above the threshold) or death due to any cause. The Kaplan-Meier method was used to estimate the distribution, and the median time to definitive 10% deterioration, along with 95% confidence intervals, was reported for each treatment group. If a patient had not had an event, time to deterioration was censored at the date of the last adequate QoL evaluation.
Time Frame: Up to approximately 29 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Months | NA [22.2 to NA] — NA = The value was not estimable due to insufficient number of participants with events | 21.2 [15.4 to 23.0]

9. Secondary Outcome: Change From Baseline in the GHS/QoL Scale Score of the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, 1 GHS/QoL scale, and 6 single items. GHS/QoL scale score ranges between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.The change from baseline in the GHS/QoL score was assessed. A positive change from baseline indicated improvement. For subjects who discontinued treatment without disease progression, post-treatment efficacy visits occurred every 8 weeks during the initial 18 months since start of treatment, followed by visits every 12 weeks until disease progression.
Time Frame: Baseline, every 2 cycles after randomization during 18 months, then every 3 cycles up to end of treatment (EOT); EOT; and every 8 or 12 weeks post-treatment until progression, assessed up to approximately 29 months. Cycle=28 days
Population: Randomized participants with data available at the specified time points. Number analyzed refers to the number of participants with an evaluable value at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 300 | 280
Score on a Scale
  Cycle 3 Day 1 | 4.6 (21.64) | 5.0 (22.10)
  Cycle 5 Day 1: number analyzed (Participants) | 277 | 246
  Cycle 5 Day 1 | 5.1 (21.81) | 5.1 (20.60)
  Cycle 7 Day 1: number analyzed (Participants) | 263 | 231
  Cycle 7 Day 1 | 5.0 (21.67) | 4.0 (22.57)
  Cycle 9 Day 1: number analyzed (Participants) | 250 | 207
  Cycle 9 Day 1 | 4.8 (22.37) | 3.7 (23.76)
  Cycle 11 Day 1: number analyzed (Participants) | 236 | 185
  Cycle 11 Day 1 | 4.3 (22.17) | 4.4 (24.53)
  Cycle 13 Day 1: number analyzed (Participants) | 213 | 166
  Cycle 13 Day 1 | 4.7 (21.14) | 3.9 (25.19)
  Cycle 15 Day 1: number analyzed (Participants) | 204 | 150
  Cycle 15 Day 1 | 4.8 (22.44) | 3.2 (24.91)
  Cycle 17 Day 1: number analyzed (Participants) | 170 | 117
  Cycle 17 Day 1 | 4.0 (20.60) | 2.7 (25.68)
  Cycle 19 Day 1: number analyzed (Participants) | 128 | 85
  Cycle 19 Day 1 | 5.5 (22.12) | -1.2 (24.10)
  Cycle 22 Day 1: number analyzed (Participants) | 79 | 46
  Cycle 22 Day 1 | 7.6 (25.43) | -3.4 (25.43)
  Cycle 25 Day 1: number analyzed (Participants) | 50 | 25
  Cycle 25 Day 1 | 5.2 (19.41) | -0.3 (25.51)
  Cycle 28 Day 1: number analyzed (Participants) | 19 | 11
  Cycle 28 Day 1 | 7.9 (19.54) | -8.3 (30.28)
  Cycle 31 Day 1: number analyzed (Participants) | 2 | 1
  Cycle 31 Day 1 | 8.3 (11.79) | -8.3
  End of treatment: number analyzed (Participants) | 129 | 179
  End of treatment | -4.4 (27.78) | -3.0 (23.41)
  Post-end of treatment 1: number analyzed (Participants) | 9 | 11
  Post-end of treatment 1 | 3.7 (25.38) | 6.8 (32.02)
  Post-end of treatment 2: number analyzed (Participants) | 3 | 2
  Post-end of treatment 2 | 5.6 (12.73) | 0.0 (11.79)
  Post-end of treatment 3: number analyzed (Participants) | 3 | 2
  Post-end of treatment 3 | 8.3 (14.43) | -4.2 (5.89)
  Post-end of treatment 4: number analyzed (Participants) | 3 | 1
  Post-end of treatment 4 | 11.1 (17.35) | -8.3
  Post-end of treatment 5: number analyzed (Participants) | 1 | 0
  Post-end of treatment 5 | 16.7 |

10. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from start of treatment to 30 days after last dose of treatment or one day before first administration of crossover treatment (for crossover participants), whichever came first.
  Crossover on-treatment deaths were collected from start of crossover treatment up to 30 days after last dose of crossover treatment.
  Post-treatment survival follow-up deaths were collected from day 31 after last dose of study treatment to end of study or one day before first administration of crossover treatment Crossover post-treatment survival follow-up deaths were collected from day 31 after last dose of crossover treatment to end of study
Time Frame: On-treatment: Up to 90 months. Crossover on-treatment: Up to approximately 33 months after crossing-over. Post-treatment survival follow-up: Up to 90 months. Crossover post-treatment survival follow-up: Up to approximately 33 months after crossing-over
Population: FAS including all randomized participants
Measure: Number; unit: Participants
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin | Placebo + NSAI/Tamoxifen+ Goserelin
Number analyzed (Participants) | 335 | 337
Participants
  On-treatment deaths | 5 | 6
  Crossover on-treatment deaths: number analyzed (Participants) | 0 | 17
  Crossover on-treatment deaths |  | 0
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 251 | 293
  Post-treatment survival follow-up deaths | 168 | 202
  Crossover post-treatment survival deaths: number analyzed (Participants) | 0 | 17
  Crossover post-treatment survival deaths |  | 1
  All deaths | 173 | 209

ADVERSE EVENTS:
Time Frame: On-treatment: from 1st dose to 30 days post-treatment or start of crossover treatment, up to 90 months Crossover on-treatment: from 1st dose of crossover treatment to 30 days post-crossover treatment, up to approximately 33 months. Post-treatment survival follow-up: from day 31 post-treatment to end of study or start of crossover treatment, up to 90 months. Crossover post-treatment survival follow-up period from day 31 post-crossover treatment to end of study, up to approximately 33 months.
Description: Safety analyses were performed in the safety set, including all participants who received at least one dose of study treatment. Deaths in the post treatment survival follow-up period are not considered Adverse Events. The total number at risk in the post-treatment survival includes patients that entered the post-treatment survival follow-up period.
Groups:
- Ribociclib + NSAI/Tamoxifen + Goserelin (On-treatment): AEs collected during on-treatment period (up to 30 days post-treatment)
- Placebo + NSAI/Tamoxifen+ Goserelin (On-treatment): AEs collected during on-treatment period (up to 30 days post-treatment or start of crossover treatment)
- Placebo Crossover to Ribociclib (On-Treatment): AEs collected during crossover on-treatment period with ribociclib for participants randomized to placebo arm who crossed-over to ribociclib (up to 30 days post- crossover treatment)
- Ribociclib + NSAI/Tamoxifen + Goserelin (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment to end of study). No AEs were collected during this period
- Placebo + NSAI/Tamoxifen+ Goserelin (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment to end of study or start of crossover treatment). No AEs were collected during this period
- Placebo Crossover to Ribociclib (Post-treatment Survival Follow-up): Deaths collected in the crossover post- treatment survival follow-up period (starting from day 31 post-crossover treatment to end of study). No AEs were collected during this period
Arm/Group | Ribociclib + NSAI/Tamoxifen + Goserelin (On-treatment) | Placebo + NSAI/Tamoxifen+ Goserelin (On-treatment) | Placebo Crossover to Ribociclib (On-Treatment) | Ribociclib + NSAI/Tamoxifen + Goserelin (Post-treatment Survival Follow-up) | Placebo + NSAI/Tamoxifen+ Goserelin (Post-treatment Survival Follow-up) | Placebo Crossover to Ribociclib (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 5/335 | 6/337 | 0/17 | 168/251 | 202/293 | 1/17
Serious Adverse Events (participants affected / at risk) | 81/335 | 49/337 | 1/17 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 326/335 | 312/337 | 14/17 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + NSAI/Tamoxifen + Goserelin (On-treatment) (N=335) | Placebo + NSAI/Tamoxifen+ Goserelin (On-treatment) (N=337) | Placebo Crossover to Ribociclib (On-Treatment) (N=17) | Ribociclib + NSAI/Tamoxifen + Goserelin (Post-treatment Survival Follow-up) (N=0) | Placebo + NSAI/Tamoxifen+ Goserelin (Post-treatment Survival Follow-up) (N=0) | Placebo Crossover to Ribociclib (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 0 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 1 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | NA | NA | NA
Axillary pain (General disorders) | 1 | 0 | 0 | NA | NA | NA
Fatigue (General disorders) | 1 | 0 | 0 | NA | NA | NA
Pyrexia (General disorders) | 4 | 4 | 0 | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | NA | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | NA | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 4 | 1 | 0 | NA | NA | NA
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | NA | NA | NA
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 2 | 0 | NA | NA | NA
COVID-19 (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Cellulitis (Infections and infestations) | 2 | 1 | 0 | NA | NA | NA
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | NA | NA | NA
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Influenza (Infections and infestations) | 2 | 1 | 0 | NA | NA | NA
Otitis media (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 5 | 1 | 0 | NA | NA | NA
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Viral infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0 | NA | NA | NA
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | NA | NA | NA
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | NA | NA | NA
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | NA | NA | NA
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
SARS-CoV-2 antibody test positive (Investigations) | 1 | 0 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | NA | NA | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | NA | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
HER2 positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | NA | NA | NA
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 1 | 1 | 0 | NA | NA | NA
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0 | NA | NA | NA
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 2 | 0 | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | NA | NA | NA
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | NA | NA | NA
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + NSAI/Tamoxifen + Goserelin (On-treatment) (N=335) | Placebo + NSAI/Tamoxifen+ Goserelin (On-treatment) (N=337) | Placebo Crossover to Ribociclib (On-Treatment) (N=17) | Ribociclib + NSAI/Tamoxifen + Goserelin (Post-treatment Survival Follow-up) (N=0) | Placebo + NSAI/Tamoxifen+ Goserelin (Post-treatment Survival Follow-up) (N=0) | Placebo Crossover to Ribociclib (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 73 | 37 | 2 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 66 | 13 | 1 | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 29 | 5 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 194 | 22 | 5 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 6 | 0 | NA | NA | NA
Lacrimation increased (Eye disorders) | 17 | 2 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 39 | 27 | 0 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 27 | 24 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 62 | 48 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 82 | 67 | 1 | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 16 | 18 | 0 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 20 | 14 | 0 | NA | NA | NA
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 113 | 78 | 4 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 48 | 30 | 0 | NA | NA | NA
Toothache (Gastrointestinal disorders) | 15 | 11 | 1 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 76 | 61 | 0 | NA | NA | NA
Asthenia (General disorders) | 54 | 43 | 1 | NA | NA | NA
Chills (General disorders) | 6 | 4 | 1 | NA | NA | NA
Fatigue (General disorders) | 89 | 86 | 2 | NA | NA | NA
Influenza like illness (General disorders) | 23 | 13 | 0 | NA | NA | NA
Localised oedema (General disorders) | 1 | 5 | 1 | NA | NA | NA
Mucosal haemorrhage (General disorders) | 0 | 0 | 1 | NA | NA | NA
Non-cardiac chest pain (General disorders) | 26 | 15 | 0 | NA | NA | NA
Oedema peripheral (General disorders) | 25 | 18 | 1 | NA | NA | NA
Pyrexia (General disorders) | 60 | 29 | 3 | NA | NA | NA
Hepatic pain (Hepatobiliary disorders) | 1 | 1 | 1 | NA | NA | NA
Contrast media reaction (Immune system disorders) | 0 | 0 | 1 | NA | NA | NA
COVID-19 (Infections and infestations) | 10 | 1 | 2 | NA | NA | NA
Herpes zoster (Infections and infestations) | 7 | 6 | 1 | NA | NA | NA
Influenza (Infections and infestations) | 29 | 24 | 1 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 34 | 23 | 0 | NA | NA | NA
Suspected COVID-19 (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 53 | 40 | 2 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 38 | 31 | 0 | NA | NA | NA
Post procedural erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 1 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 58 | 34 | 2 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 55 | 36 | 4 | NA | NA | NA
Blood cholesterol increased (Investigations) | 12 | 9 | 1 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 42 | 16 | 1 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 22 | 32 | 0 | NA | NA | NA
Neutrophil count decreased (Investigations) | 119 | 5 | 4 | NA | NA | NA
SARS-CoV-2 test negative (Investigations) | 2 | 0 | 1 | NA | NA | NA
SARS-CoV-2 test positive (Investigations) | 5 | 1 | 1 | NA | NA | NA
Weight increased (Investigations) | 9 | 10 | 1 | NA | NA | NA
White blood cell count decreased (Investigations) | 55 | 4 | 1 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 34 | 27 | 1 | NA | NA | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 15 | 13 | 1 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 18 | 0 | NA | NA | NA
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 | 17 | 2 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 130 | 122 | 1 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 76 | 72 | 0 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 34 | 32 | 0 | NA | NA | NA
Joint stiffness (Musculoskeletal and connective tissue disorders) | 11 | 12 | 1 | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 10 | 0 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 | 20 | 0 | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 17 | 0 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 42 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 19 | 19 | 0 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 53 | 44 | 0 | NA | NA | NA
Ageusia (Nervous system disorders) | 3 | 0 | 1 | NA | NA | NA
Dizziness (Nervous system disorders) | 27 | 25 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 96 | 89 | 1 | NA | NA | NA
Loss of consciousness (Nervous system disorders) | 1 | 2 | 1 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 18 | 18 | 0 | NA | NA | NA
Syncope (Nervous system disorders) | 2 | 4 | 1 | NA | NA | NA
Anxiety (Psychiatric disorders) | 22 | 17 | 0 | NA | NA | NA
Depression (Psychiatric disorders) | 22 | 23 | 0 | NA | NA | NA
Insomnia (Psychiatric disorders) | 51 | 55 | 0 | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 24 | 23 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 42 | 3 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 21 | 1 | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 33 | 18 | 0 | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 | 13 | 0 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 64 | 41 | 2 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 8 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 39 | 18 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 53 | 32 | 0 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 1 | 1 | NA | NA | NA
Hot flush (Vascular disorders) | 118 | 117 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 42 | 28 | 0 | NA | NA | NA
Lymphoedema (Vascular disorders) | 8 | 11 | 1 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT02278120/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT02278120/SAP_003.pdf